CLINICAL TRIAL: NCT03127826
Title: Validation of the STarT Back Screening Tool in the Primary Care Management of Low Back Pain in the Military Health System: A Randomized Trial of Risk-stratified vs. Usual Care
Brief Title: Validation of the STarT Back Screening Tool in the Military
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brooke Army Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Dan Rhon, Director of Clinical Outcomes Research at the Center for the Intrepid, Brooke Army Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C.2016.047d
Record Dates: First submitted 2017-04-14; First posted 2017-04-25 (Actual); Last update posted 2022-06-01 (Actual); Status verified 2022-05

CONDITIONS: Low Back Pain; Lumbago; Radiculopathy; Intervertebral Disc Disorder
Keywords: Low Back Pain; Risk-Stratified Care
MeSH Terms: conditions — Low Back Pain; Radiculopathy; Intervertebral disc disease

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Masking Description: Primary care providers will be unaware of risk stratification scores.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (Active Comparator): * "Managing Low Back Pain" pamphlet from DoD/VA
  * No specific guidance regarding physical therapy (PT) or other referrals, thus decision to refer or not will be made by the primary care manager (PCM) according to their preference
  Interventions: Procedure: Usual Care
- Risk Stratified Care (Experimental): * "Managing Low Back Pain" pamphlet from DoD/VA
  * Self-management education and tools
  * 2-item spinal manipulation screening/delivery if indicated
  Low Risk:
  * Home Exercise Program as indicated
  * No referral for ongoing physical therapy
  Medium Risk and High Risk
  * Referral to physical therapy for ongoing care at physical therapists discretion
  * Managed by a "psychologically informed physical therapy" trained physical therapist
  Interventions: Procedure: Risk Stratified Care

INTERVENTIONS:
Procedure: Risk Stratified Care — Physical therapists providing care will all have attended live training in PIPT principles and be involved in monthly continuing education on these principles. The use of specific principles is guided by the patient's risk stratification (as determined by the STarT Back Tool).
  Medium Risk:
  - Reassurance will be provided to address specific concerns related to their LBP and implications on work
  High Risk:
  - Physical therapy will be psychologically augmented with the assessment of biopsychosocial risk factors and the adoption of cognitive behavioral principles that explore patient concerns and address unhelpful beliefs and behaviors, including tailored education (e.g., stress management and pain neuroscience), graded exercise, & graded exposure
  Arms: Risk Stratified Care
Procedure: Usual Care — Usual care at the general practitioner's discretion
  Arms: Usual Care

SUMMARY:
This is a trial to validate the use of the STarT Back Screening Tool (SBST) in the Military Health System for patients with low back pain presenting to primary care.

DETAILED DESCRIPTION:
Subjects with low back pain presenting to primary care will be enrolled in a study that aims to evaluate the utility of the SBST for providing risk-stratified care. The concept of this approach revolves around matching treatment to patients based on their risk for developing chronic disability from back pain. Those at low risk receive less treatment, and those at high risk need more specialized treatment, that includes psychosocially-focused and cognitive considerations. This approach will be compared to usual care, where general practitioners carry out the course of action they think best for each patient, without any other guidance. Patients will be followed for 1 year.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females who are between the ages of 18-50 years old
2. Primary complaint of LBP for any duration, with or without associated radiculopathy
3. Can speak and understand English
4. Be willing and able to give full, informed written consent

Exclusion Criteria:

1. Red Flags: Any potentially serious or systemic disorders (e.g., cauda equina compression, inflammatory arthritis, compression fracture, malignancy, infection, severe neurological progression), serious illness or comorbidity
2. Spinal surgery in the past 24 months
3. Current pregnancy (or within the last 6 months)
4. Already receiving treatment (other than primary care) for this episode of LBP
5. Inability to attend regular treatment sessions
6. Pending litigation or a medical evaluation board

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 290 (Actual)
Dates: Start 2017-04-07 (Actual); Primary Completion 2021-02-26 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
Roland-Morris Disability Questionnaire (RMDQ) | 1 year
  The focus of the interventions is directed towards the secondary prevention of disabling back pain. The RMDQ will be used to assess physical disability. The RMDQ is a recommended disability measure that it is widely used in LBP studies in primary care and was the primary outcome used in the STarT Back trial by Hill et al. (2011). The form provides 24 statements and prompts the participant by stating "When your back hurts, you may find it difficult to do some of the things you normally do." Then it states, "Mark only the sentences that describe you today." Examples include "I avoid heavy jobs around the house because of my back" and "I find it difficult to turn over in bed because of my back". Scores are calculated by percent improvement from baseline to post-intervention [(points of improvement made/total items checked at baseline) x 100]

SECONDARY OUTCOMES:
Patient Acceptable Symptom Scale (PASS) | 1 year
  Often defined as "the highest level of symptoms beyond which patients consider themselves well." This outcome measure has been used in previous studies looking at the effects of cervical thoracic thrust manipulation on shoulder pain. The question that will be asked to assess this level is, "Taking into account all the activities you have during your daily life, your level of pain, and also your functional impairment, do you consider that your current state is satisfactory?" Individuals who respond "yes" will be categorized as a success."
Credibility Expectancy Questionnaire (CEQ) | 1 year
  The CEQ is a 6-item self-report measure evaluating treatment credibility and expectations for improvement. This will be assessed at baseline after treatment group assignment is revealed to provide descriptive information about participants' perceptions of their treatment assignment and optimism for improvement. The CEQ may be used as a covariate if perceptions differ meaningfully between groups as participants' initial perceptions of treatment credibility can impact outcomes.
Patient Reported Outcomes Measurement Information System 57-Item Profile v 2.0 (PROMIS-57) | 1 year
  The PROMIS 57 efficiently assesses several outcomes important to patients including pain intensity and interference, sleep disturbance, anxiety, depression, fatigue, and social role participation using items developed with rigorous methodology and patient input. This is a 57-item questionnaire with 8 questions per domain.
EuroQoL (EQ-5D) | 1 year
  The EQ-5D is a generic quality of life questionnaire that will assess quality of life on a scale that can be referenced to other disease conditions. The EQ-5D covers 5 domains: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each domain has 3 response categories: level 1, "no problems"; level 2, "some problems"; and level 3, "inability or extreme problems." Responses are combined to give a 5-digit descriptive health state classification (e.g., 11222). The EQ-5D yields a total of 243 possible health states. Valuations for each health state are available. The EQ-5D is commonly used in economic evaluation of interventions and cost-effectiveness analysis.
Healthcare Utilization | 2 years
  Low back pain related healthcare costs

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Rhon, DPT, DSc, Principal Investigator — Director of Clinical Outcomes Research, Center for the Intrepid
Locations (1):
- Brooke Army Medical Center, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Data sharing must go through a Data Sharing Agreement via the Defense Health Agency
Time Frame: Usually the Data Sharing Agreement with the Defense Health Agency is good for 1 year. But the terms are all unique and contract-specific.
Access Criteria: Through a proper Data Sharing Agreement Application (DSAA) with the US Defense Health Agency
URL: https://www.health.mil/Military-Health-Topics/Privacy-and-Civil-Liberties/Submit-a-Data-Sharing-Application

REFERENCES:
- [Background] Hill JC, Whitehurst DG, Lewis M, Bryan S, Dunn KM, Foster NE, Konstantinou K, Main CJ, Mason E, Somerville S, Sowden G, Vohora K, Hay EM. Comparison of stratified primary care management for low back pain with current best practice (STarT Back): a randomised controlled trial. Lancet. 2011 Oct 29;378(9802):1560-71. doi: 10.1016/S0140-6736(11)60937-9. Epub 2011 Sep 28. PMID 21963002
- [Background] Beneciuk JM, Fritz JM, George SZ. The STarT Back Screening Tool for prediction of 6-month clinical outcomes: relevance of change patterns in outpatient physical therapy settings. J Orthop Sports Phys Ther. 2014 Sep;44(9):656-64. doi: 10.2519/jospt.2014.5178. Epub 2014 Aug 6. PMID 25098194
- [Background] Main CJ, Sowden G, Hill JC, Watson PJ, Hay EM. Integrating physical and psychological approaches to treatment in low back pain: the development and content of the STarT Back trial's 'high-risk' intervention (StarT Back; ISRCTN 37113406). Physiotherapy. 2012 Jun;98(2):110-6. doi: 10.1016/j.physio.2011.03.003. Epub 2011 Jun 12. PMID 22507360
- [Background] Beneciuk JM, George SZ. Pragmatic Implementation of a Stratified Primary Care Model for Low Back Pain Management in Outpatient Physical Therapy Settings: Two-Phase, Sequential Preliminary Study. Phys Ther. 2015 Aug;95(8):1120-34. doi: 10.2522/ptj.20140418. Epub 2015 Apr 9. PMID 25858972
- [Background] Saunders B, Bartlam B, Foster NE, Hill JC, Cooper V, Protheroe J. General Practitioners' and patients' perceptions towards stratified care: a theory informed investigation. BMC Fam Pract. 2016 Aug 31;17(1):125. doi: 10.1186/s12875-016-0511-2. PMID 27582134
- [Derived] Rhon DI, Greenlee TA, Poehlein E, Beneciuk JM, Green CL, Hando BR, Childs JD, George SZ. Effect of Risk-Stratified Care on Disability Among Adults With Low Back Pain Treated in the Military Health System: A Randomized Clinical Trial. JAMA Netw Open. 2023 Jul 3;6(7):e2321929. doi: 10.1001/jamanetworkopen.2023.21929. PMID 37410465